CLINICAL TRIAL: NCT06649799
Title: Comparative Study on Changes in Anterior Chamber Cytokines, Oxidative Stress, and Pupil Size After LenSx and Z8 Femtosecond Lasers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022-0672
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Cataract
Keywords: cataract; femtosecond laser; cytokines; oxidative stress; miosis;
MeSH Terms: conditions — Cataract; Miosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LenSx (Experimental)
  Interventions: Device: LenSx
- Z8 (Placebo Comparator)
  Interventions: Device: Z8

INTERVENTIONS:
Device: LenSx — The patients in Group 1 conduct FLACS under LenSx
  Arms: LenSx
Device: Z8 — The patients in Group 1 conducted FLACS using Z8
  Arms: Z8

SUMMARY:
Femtosecond laser-assisted cataract surgery is rapidly gaining popularity. Among the 5 femtosecond laser platforms available at present for cataract surgery, the Femto LDV Z8 (Ziemer Ophthalmic Systems AG) is a high-frequency system and delivers energy pulses in nanojoule levels, while Lensx platform (Lensx, Alcon Laboratories, Inc.) used a high-energy laser system. In femtosecond laser-assisted cataract surgery, the laser pretreatment is associated with breakdown of blood-aqueous barrier (BAB) associated with increased aqueous total prostaglandin, cytokines and Oxygen-free radicals concentration. The prostaglandin rise immediately after laser pretreatment is further thought to be the causative factor for the intraoperative miosis in femtosecond laser-assisted cataract surgery. However, the analysis of anterior chamber inflammatory factors, oxidative stress, and pupil size after femtosecond laser-assisted cataract surgery between different laser platforms has not been investigated in clinical studies. Understanding the cytokine and chemokine changes related to the laser pretreatment provides better insight into the inflammatory response in femtosecond laser-assisted cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

Age related cataracts over 50 years old, nuclear grades II-III

Exclusion Criteria:

* Eye diseases: glaucoma, uveitis

  * Systemic diseases: autoimmune diseases such as diabetes and rheumatism ③ Intraoperative complications: ④ Medication history: Over 1 month before surgery, systemic or local hormones, NASIDs ⑤ History of eye surgery (including YAG laser and fundus laser), trauma

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
PGE2 | through study completion, an average of half a year
  The concentrations of PGE2 in aqueous humor
cytokines (IL-1β、IL-6, IL-8、TNF-a) | through study completion, an average of half a year
  The concentrations of cytokines (IL-1β、IL-6, IL-8、TNF-a) in aqueous humor
MDA | through study completion, an average of half a year
  The concentrations of MDA in aqueous humor

SECONDARY OUTCOMES:
central corneal thickness | through study completion, an average of half a year
  The central corneal thickness was measured
central macular thickness | through study completion, an average of half a year
  The central macular thickness was measured

CONTACTS AND LOCATIONS:
Locations (1):
- ye Center, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No